CLINICAL TRIAL: NCT02402816
Title: MPP Narrow QRS:Pilot Study on Multipoint Pacing in Patients With Narrow QRS
Brief Title: MPP Narrow QRS:Pilot Study on Multipoint Pacing in Patients With QRS Beetwen 100 and 130 Msec
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Humanitas Hospital, Italy (Other)
Responsible Party: Principal Investigator, Dr.Maurizio Gasparini, MD, Humanitas Hospital, Italy
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1.0
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Defibrillators, Implantable

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MPP ON (Experimental): Patients will be randomized to the MPP-ON Arm vs Standard ICD
  Interventions: Device: MultiPoint Pacing ON
- Standard ICD (Active Comparator): Patients will be randomized to the MPP-ON Arm vs Standard ICD
  Interventions: Device: Implantable cardioverter-defibrillator (ICD)

INTERVENTIONS:
Device: MultiPoint Pacing ON — MultiPoint Pacing ON
  Arms: MPP ON
Device: Implantable cardioverter-defibrillator (ICD) — Implantable cardioverter-defibrillator (ICD)
  Arms: Standard ICD

SUMMARY:
The purpose of this study is to assess the impact of the Multi Point Pacing (MPP) feature in the treatment of patients with QRS beetwen 100 and 130 msec in patients candidate to ICD implant.

ELIGIBILITY:
Inclusion Criteria:

* Patients with EF < 35% on OPT at least 3 months and candidate to ICD
* QRS duration: 100-130 ms
* Patients willing and able to comply with study requirements
* Must indicate their understanding of the study and willingness to participate by signing an appropriate informed consent form
* Successful quadripolar LV lead implant (only for Treatment Group)

Exclusion Criteria:

* Myocardial Infarction, unstable angina within 40 days prior the enrollment
* Patients with no left ventricular contractile reserve after low dose dobutamine stress echocardiography test
* Recent cardiac revascularization (PTCA, Stent or CABG) in the 4 weeks prior to enrollment or planned for the 3 months following
* Cerebrovascular Accident (CVA) or Transient Ischemic Attack (TIA) in the 3 months prior the enrollment
* Primary valvular disease
* Unable to comply with the follow up schedule
* Less than 18 years of age
* Pregnant or are planning to become pregnant during the duration of the investigation
* Classification of Status 1 for cardiac transplantation or consideration for transplantation over the next 12 months
* Undergone a cardiac transplantation
* Life expectancy < 12 months
* Patients with permanent Atrial fibrillation
* Patients with Nyha 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients presenting reverse remodeling (reduction of ESV > 15%) after 6 and 12 months | up to 12 Months

SECONDARY OUTCOMES:
Percentage of patients presenting reverse remodeling (reduction of ESV > 15%) after 24 months | 24-Months
Percentage of responder patients in term of increase of EF > 5 points % at 12 months Follow-Up | 12-Months
Percentage of responder patients in term of increase of EF > 5 points % at 24 months Follow-Up | 24-Months
Percentage of responder patients in term of BNP < 400 pg/ml at 12 months | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Gasparini, MD, Principal Investigator — Humanitas Research Hospital-Rozzano-Italy
Locations (6):
- Italy (6):
  - Ospedale Maggiore di Crema, Crema
  - A.O. Niguarda Ca' Granda, Milan
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Ospedale S.Maria della Misericordia, Rovigo
  - Humanitas Research Hospital, Rozzano
  - Ospedale Santa Maria della Misericordia, Udine

REFERENCES:
- [Derived] Gasparini M, Galimberti P, Bragato R, Ghio S, Raineri C, Landolina M, Chieffo E, Lunati M, Mulargia E, Proclemer A, Facchin D, Rordorf R, Vicentini A, Marcantoni L, Zanon F, Klersy C. Multipoint Pacing versus conventional ICD in Patients with a Narrow QRS complex (MPP Narrow QRS trial): study protocol for a pilot randomized controlled trial. Trials. 2016 Dec 3;17(1):572. doi: 10.1186/s13063-016-1698-1. PMID 27927248